CLINICAL TRIAL: NCT00983190
Title: HeartMate II BeneMACS Long Term LVAD Study
Brief Title: BeneMACS Study:HeartMate 2 (HM2)Left Ventricular Assist Device (LVAD) Survival in Non Transplant Patients is Equal/Better Than Results in Medical Literature
Acronym: BeneMACs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Collaborators: KU Leuven (Other); Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other); Interagency Registry for Mechanical Assisted Circulatory Support (INTERMACS) (Unknown); Thoratec Corporation (Industry); Thoratec Europe Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BeneMACS LVAD Study Rev 6Jan09; B32220096329 - Belgium
Record Dates: First submitted 2009-09-22; First posted 2009-09-24 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Heart Failure
Keywords: HeartMate II; BeneMACS; LVAD; Thoratec Corporation
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Group Assignment (Other)
  Interventions: Device: Left Ventricular Assist Device (HeartMate II)

INTERVENTIONS:
Device: Left Ventricular Assist Device (HeartMate II) — The HM II is a high speed, electric, axial flow, rotary blood pump. The pump drains blood from the left ventricular apex via rigid inlet cannulae and ejects into the aortic root via an outflow cannula joined to the aorta with an end to side anastamosis. Power and control of the pump are delivered through a percutaneous cable from pump to the belt-worn System Controller. The System Controller will receive power from the Power Base Unit (PBU), or two battery modules that may be worn in shoulder holsters or on the belt
  Other Names: HeartMate II; LVAD; HMII

SUMMARY:
Study Purpose

The purpose of the BeneMACS Long-Term LVAD Study is to demonstrate that survival in non transplant patients implanted with the HeartMate II LVAD as destination therapy in Belgium and the Netherlands are equivalent to or better than published results in the scientific literature with approved devices. Implants will be performed following the HeartMate II guidelines.

Characterization of Patient Population The HeartMate II will be implanted as destination therapy in patients who are not candidates for cardiac transplantation.

Study Design

The study is a prospective, non-randomized, non-blinded multi-center study with historical control. The study will consist of the assignment of eligible patients to treatment with the LVAD. The first 10 patients to have the device implanted will be enrolled in the study.

Study End point

Patients enrolled in the study will be followed until end points defined as death, 2-year support on the HeartMate II, device removal, transplantation, or recovery.

Data Collection and Follow-up

All data will be entered into INTERMACS® through their web-based data entry system. All data for the BeneMACs study will be held separately from the main INTERMACS database, and used only for the purpose of the BeneMACs study.

Investigator sites

Cliniques Universitaires St. Luc, Avenue Hippocrates 10, 1200 Brussels, Belgium Leuven Gasthuisberg University Hospital, Herestraat 49, 3000 Leuven, Belgium

DETAILED DESCRIPTION:
1. STUDY OBJECTIVE

   The purpose of the BeneMACs Long-Term LVAD Study is to demonstrate that survival in non transplant patients implanted with the HeartMate II LVAD as destination therapy in Belgium and the Netherlands are equivalent to or better than published results in the scientific literature with approved devices. (see section 4.6.4) Implants will be performed following the HeartMate II guidelines.
2. STUDY ENTRY CRITERIA - PATIENT SELECTION

   2.1 Characterization of Patient Population The HeartMate II will be implanted as destination therapy in patients who are not candidates for cardiac transplantation.
3. METHODS

3.1 Study Design

The study is a prospective, non-randomized, non-blinded multi-center study with historical control. The study will consist of the assignment of eligible patients to treatment with the LVAD. The first 10 patients to have the device implanted will be enrolled in the study.

3.2 Study End point

Patients enrolled in the study will be followed until end points defined as death, 2-year support on the HeartMate II, device removal, transplantation, or recovery.

3.3 Number of Clinical Sites and Patients

The study will be conducted at up to three (3) clinical sites. A total of 10 patients (3-4 patients per site) will be enrolled and implanted with the HM II.

3.4 Data Collection and Follow-up:

All data will be entered into INTERMACS® through their web-based data entry system. Complete documentation and the Site User's Guide are contained at the data entry website (www.intermacs.org). INTERMACS (the Interagency Registry of Mechanical Assisted Circulatory Support) was formed as a partnership between the National Heart Lung, and Blood Institute (NHLBI), the FDA, Centers for Medicare and Medicaid Services (CMS), participating hospitals and industry (reference 7.2). It is the main MCS registry in the United States. In addition to its primary purpose, the validated database used by INTERMACS is also being made available as a service to other studies of mechanical circulatory support devices such as the BeneMACs study.

All data for the BeneMACs study will be held separately from the main INTERMACS database, and used only for the purpose of the BeneMACs study.

ELIGIBILITY:
Inclusion Criteria:

* Patient or their legal representative has signed an informed consent. > 18 years of age.
* BSA > 1.3m2.
* Patients with advanced heart failure symptoms (Class IIIB or IV) who are: (patient must meet one of the following) On optimal medical management, including dietary salt restriction, diuretics, beta-blockers, spironolactone and ACE inhibitors, for at least 45 out of the last 60 days and are failing to respond; or In Class III or Class IV heart failure for at least 14 days, and dependent on intra aortic balloon pump (IABP) for 5 days and/or inotropes for at least 10 days; or Treated with ACE inhibitors or beta-blockers for at least 30 days and found to be intolerant.
* Female patients of childbearing potential must agree to use adequate contraceptive precautions (defined as oral contraceptives, intrauterine devices, surgical contraceptives or a combination of condom and spermicide) for the duration of the study.
* Ineligible for cardiac transplant.
* VO2max < 14 ml/kg/min or <50% of predicted VO2max with attainment of anaerobic threshold (AT), if not contra-indicated due to IV inotropes, angina or physical disability.
* LVEF is < 25%.

Exclusion Criteria:

* Etiology of heart failure is due to or associated with uncorrected thyroid disease, obstructive cardiomyopathy, pericardial disease, amyloidosis, active myocarditis or restrictive cardiomyopathy.
* Technical obstacles, which pose an inordinately high surgical risk, in the judgment of the investigator.
* Body Mass Index (BMI) > 40 kg/m2.
* Positive pregnancy test if female of childbearing age.
* Presence of mechanical aortic valve that will not be converted to a bioprosthesis at time of LVAD implant.
* History of cardiac transplant or cardiomyoplasty.
* Platelet count < 50,000.
* Evidence of an untreated aortic aneurysm > 5cm.
* Psychiatric disease, irreversible cognitive dysfunction or psychosocial issues that are likely to impair compliance with the study protocol and LVAD management.
* Presence of active, uncontrolled infection.
* Intolerance to anticoagulant or antiplatelet therapies or any other peri/post operative therapy the investigator will require based upon the patient's health status.
* INR > 2.5, which is not due to anti-coagulant therapy, or Plavix administration within 5 days.
* Evidence of intrinsic hepatic disease as defined by liver enzyme values (AST or ALT or total bilirubin) that are > 5 times the upper limit of normal, or biopsy proven liver cirrhosis.
* History of severe COPD or severe restrictive lung disease.
* Fixed pulmonary hypertension with a PVR > 8 Wood units that is unresponsive to pharmacological intervention.
* History of a stroke within 90 days prior to enrollment, or a history of cerebral vascular disease with significant (> 80%) extra cranial stenosis.
* Serum creatinine > 3.5 mg/dl or the need for chronic renal replacement therapy (e.g. chronic dialysis).
* Significant peripheral vascular disease accompanied by rest pain or extremity ulceration.
* The patient has moderate to severe aortic insufficiency without plans for correction during pump implantation surgery.
* Participation in any other clinical investigation that is likely to confound study results or affect study outcome.
* Any condition, other than heart failure, that is likely to limit survival to less than 3 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-07; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Study will assign patients to treatment with an HMII LVAD. Ten patients will be enrolled in the study. Patients enrolled in the study will be followed until end points defined as 2year support on device, device removal, transplantation recovery, or death | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bart Meyns, MD/PhD, Principal Investigator — Leuven Gasthuisberg University Hospital; Luc-Marie Jacquet, MD/PhD, Principal Investigator — Cliniques Universitaires St Luc
Locations (2):
- Belgium (2):
  - Cliniques Universitaires St Luc, Brussels
  - Leuven Gasthuisberg University Hospital, Leuven